CLINICAL TRIAL: NCT00378508
Title: Phase II Trial of hOKT3gamma1(Ala-Ala) Teplizumab for Treatment of Patients With Recent Onset Type 1 Diabetes
Brief Title: Anti-CD3 mAb Treatment of Recent Onset Type 1 Diabetes
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH); Juvenile Diabetes Research Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Delay-Study 5; R01DK057846 (NIH)
Record Dates: First submitted 2006-09-18; First posted 2006-09-20 (Estimated); Results first posted 2012-10-31 (Estimated); Last update posted 2021-08-13 (Actual); Status verified 2021-08

CONDITIONS: Type 1 Diabetes Mellitus
Keywords: immune therapy; autoimmunity; insulin secretion; diabetes mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Autoimmune Diseases; Diabetes Mellitus | interventions — teplizumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): The course of Teplizumab comprises daily doses of 51 µg/m2, 103 µg/m2, 207 µg/m2, 413 µg/m2, and 10 of 826 µg/m2 over a 14 day treatment period.
  Interventions: Drug: mAb hOKT3gamma1(Ala-Ala), Teplizumab
- 2 (Placebo Comparator): Normal saline infusion
  Interventions: Drug: Placebo Arm

INTERVENTIONS:
Drug: mAb hOKT3gamma1(Ala-Ala), Teplizumab — This is a randomized, two-arm, double blind placebo controlled phase II trial in which 60 participants with recent-onset T1DM are randomized at a 1:1 ratio to receive Teplizumab or placebo over a 14 day treatment period. The course of Teplizumab comprises daily doses of 51 µg/m2, 103 µg/m2, 207 µg/m2, 413 µg/m2, and 10 of 826 µg/m2.
  Other Names: mAb hOKT3gamma1(Ala-Ala), MGA031, Teplizumab
  Arms: 1
Drug: Placebo Arm
  Arms: 2

SUMMARY:
This is a randomized placebo controlled study to test whether a single 14 course of treatment with the anti-CD3 monoclonal antibody, hOKT3gamma1(Ala-Ala),Teplizumab will prevent the loss of insulin secretory capacity in individuals with Type 1 diabetes of 4 - 12 months duration since diagnosis.

DETAILED DESCRIPTION:
The study design is a double blind placebo controlled trial that will enroll subjects between the ages of 8 - 30 who have had the diagnosis of Type 1 diabetes made 4 - 12 months prior to enrollment. A single 14 course of treatment with mAb hOKT3gamma1(Ala-Ala), Teplizumab will be given. The primary endpoint is the C-peptide response to a mixed meal at 12 months. A total of 60 subjects will be enrolled (30 in the drug treatment and 30 in the placebo groups) at 4 study sites: Yale University,the University of California at San Francisco, Children's Hospital of Philadelphia, and the Barbara Davis Diabetes Center.

ELIGIBILITY:
Inclusion Criteria:

* age 8 - 30,
* duration of diabetes 4 - 12 months,
* weight greater than 27.5 kg,
* stimulated C-peptide >= 0.2 pmol/ml

Exclusion Criteria:

* asthma,
* history of hepatitis C, hepatitis B, HIV

Ages: 8 Years to 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 63 (Actual)
Dates: Start 2006-09; Primary Completion 2011-08 (Actual); Study Completion 2013-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kevan C Herold, Principal Investigator — Yale University; Jeffrey A Bluestone, PhD, Principal Investigator — University of California at San Francisco
Locations (4):
- United States (4):
  - University of California at San Francisco, San Francisco, California
  - Barbara Davis Diabetes Center, Aurora, Colorado
  - Yale University, New Haven, Connecticut
  - Children's Hospital of Philadelphia (CHOP), Philadelphia, Pennsylvania

REFERENCES:
- [Background] Herold KC, Hagopian W, Auger JA, Poumian-Ruiz E, Taylor L, Donaldson D, Gitelman SE, Harlan DM, Xu D, Zivin RA, Bluestone JA. Anti-CD3 monoclonal antibody in new-onset type 1 diabetes mellitus. N Engl J Med. 2002 May 30;346(22):1692-8. doi: 10.1056/NEJMoa012864. PMID 12037148
- [Background] Herold KC, Gitelman SE, Masharani U, Hagopian W, Bisikirska B, Donaldson D, Rother K, Diamond B, Harlan DM, Bluestone JA. A single course of anti-CD3 monoclonal antibody hOKT3gamma1(Ala-Ala) results in improvement in C-peptide responses and clinical parameters for at least 2 years after onset of type 1 diabetes. Diabetes. 2005 Jun;54(6):1763-9. doi: 10.2337/diabetes.54.6.1763. PMID 15919798
- [Derived] Sherr JL, Ghazi T, Wurtz A, Rink L, Herold KC. Characterization of residual beta cell function in long-standing type 1 diabetes. Diabetes Metab Res Rev. 2014 Feb;30(2):154-62. doi: 10.1002/dmrr.2478. PMID 24115337
- [Derived] Lebastchi J, Deng S, Lebastchi AH, Beshar I, Gitelman S, Willi S, Gottlieb P, Akirav EM, Bluestone JA, Herold KC. Immune therapy and beta-cell death in type 1 diabetes. Diabetes. 2013 May;62(5):1676-80. doi: 10.2337/db12-1207. Epub 2013 Feb 19. PMID 23423576
- [Derived] Herold KC, Gitelman SE, Willi SM, Gottlieb PA, Waldron-Lynch F, Devine L, Sherr J, Rosenthal SM, Adi S, Jalaludin MY, Michels AW, Dziura J, Bluestone JA. Teplizumab treatment may improve C-peptide responses in participants with type 1 diabetes after the new-onset period: a randomised controlled trial. Diabetologia. 2013 Feb;56(2):391-400. doi: 10.1007/s00125-012-2753-4. Epub 2012 Oct 21. PMID 23086558

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were recruited from 4 clinical sites and were eligible if they were between the ages of 8-30 and diagnosed with Type 1 Diabetes for at least 4 months, but not more than 12 months prior to enrollment.
Groups:
- Saline Infusions (Placebo): The course of normal saline infusion comprises daily doses of 51 µg/m2, 103 µg/m2, 207 µg/m2, 413 µg/m2, and 10 of 826 µg/m2 over a 14 day treatment period.
- Teplizumab Infusion (Active): The course of teplizumab infusion comprises daily doses of 51 µg/m2, 103 µg/m2, 207 µg/m2, 413 µg/m2, and 10 of 826 µg/m2 over a 14 day treatment period.
Period: Overall Study
Arm/Group | Saline Infusions (Placebo) | Teplizumab Infusion (Active)
Started | 29 | 34
Randomized | 29 | 34
Received Intervention/Placebo | 28 | 31
Completed | 27 | 31
Not Completed | 2 | 3
Not completed — Withdrawal by Subject | 1 | 3
Not completed — Lost to Follow-up | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Teplizumab Infusions (Active): The course of teplizumab infusion comprises daily doses of 51 µg/m2, 103 µg/m2, 207 µg/m2, 413 µg/m2, and 10 of 826 µg/m2 over a 14 day treatment period.
- Total: Total of all reporting groups
Arm/Group | Saline Infusions (Placebo) | Teplizumab Infusions (Active) | Total
Number analyzed (Participants) | 27 | 31 | 58
Age, Customized [Number; unit: participants]
  <15 years | 20 | 18 | 38
  >=15 years | 7 | 13 | 20
Sex/Gender, Customized [Number; unit: participants]
  Female | 10 | 15 | 25
  Male | 17 | 16 | 33

OUTCOME MEASURES:

1. Primary Outcome: C-peptide Area Under the Curve (AUC) Response to a Mixed Meal Tolerance Test (MMTT) at 12 Months
Description: C-peptide secretory response was calculated as ln[(Area Under the Curve of the C-peptide from the 240 minute MMTT/240 +1]
  For presentation, the C-peptide data were converted to the AUC as pmol/ml. This is adjusted for baseline.
Time Frame: At month 12 post-treatment
Population: This endpoint was compared in the modified intent to treat population which included all subjects with at least one post-randomization mixed meal tolerance test (MMTT)
Measure: Least Squares Mean (95% Confidence Interval); unit: pmol/ml
Arm/Group | Teplizumab Infusions (Active) | Saline Infusions (Placebo)
Number analyzed (Participants) | 31 | 27
pmol/ml | 0.451 [0.4 to 0.505] | 0.371 [0.319 to 0.424]

2. Secondary Outcome: Hemoglobin A1c
Time Frame: At 12 months post-treatment
Measure: Least Squares Mean (95% Confidence Interval); unit: percentage of hemogloblin A1c
Arm/Group | Teplizumab Infusions (Active) | Saline Infusions (Placebo)
Number analyzed (Participants) | 31 | 27
percentage of hemogloblin A1c | 6.85 [6.47 to 7.23] | 7.35 [6.87 to 7.83]

3. Secondary Outcome: Average Insulin Use Over 12 Months
Time Frame: After 12 months post-treatment
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: U/kg/d
Groups:
- Saline Infusion (Placebo): The course of normal saline infusion comprises daily doses of 51 µg/m2, 103 µg/m2, 207 µg/m2, 413 µg/m2, and 10 of 826 µg/m2 over a 14 day treatment period.
Arm/Group | Teplizumab Infusions (Active) | Saline Infusion (Placebo)
Number analyzed (Participants) | 31 | 27
U/kg/d | 0.475 [0.428 to 0.521] | 0.574 [0.0526 to 0.622]

4. Primary Outcome: C-peptide Area Under the Curve (AUC) Response to a Mixed Meal Tolerance Test (MMTT) at Baseline
Description: C-peptide secretory response was calculated as ln[(Area Under the Curve of the C-peptide from the 240 minute MMTT/240 +1]
  For presentation, the C-peptide data were converted to the AUC as pmol/ml. This baseline data was used to adjust for the C-peptide AUC primary endpoint measure at 12 months.
Time Frame: At Baseline (before treatment)
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: pmol/ml
Arm/Group | Teplizumab Infusions (Active) | Saline Infusions (Placebo)
Number analyzed (Participants) | 31 | 27
pmol/ml | 0.593 [0.493 to 0.699] | 0.554 [0.417 to 0.705]

5. Secondary Outcome: Baseline Insulin Use
Time Frame: At baseline (before treatment)
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: U/kg/d
Arm/Group | Teplizumab Infusions (Active) | Saline Infusion (Placebo)
Number analyzed (Participants) | 31 | 27
U/kg/d | 0.405 [0.354 to 0.456] | 0.386 [0.308 to 0.464]

6. Secondary Outcome: Baseline Hemoglobin A1c
Time Frame: At baseline (before treatment)
Measure: Least Squares Mean (95% Confidence Interval); unit: percentage of hemoglobin A1c
Arm/Group | Teplizumab Infusions (Active) | Saline Infusions (Placebo)
Number analyzed (Participants) | 31 | 27
percentage of hemoglobin A1c | 6.32 [6.04 to 6.60] | 7.1 [6.66 to 7.64]

ADVERSE EVENTS:
Time Frame: The adverse event data was collected throughout the duration of the study which was approximately 6 years.
Groups:
- Saline Infusions (Placebo): The course of a saline infusion comprises daily doses of 51 µg/m2, 103 µg/m2, 207 µg/m2, 413 µg/m2, and 10 of 826 µg/m2 over a 14 day treatment period.
Arm/Group | Saline Infusions (Placebo) | Teplizumab Infusion (Active)
Serious Adverse Events (participants affected / at risk) | 0/29 | 1/34
Other Adverse Events (participants affected / at risk) | 29/29 | 25/34
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs:
Term (organ system) | Saline Infusions (Placebo) (N=29) | Teplizumab Infusion (Active) (N=34)
Drug Related Hypersensitivity (Immune system disorders) | 0 | 1/33
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs:
Term (organ system) | Saline Infusions (Placebo) (N=29) | Teplizumab Infusion (Active) (N=34)
Abdominal Discomfort (Gastrointestinal disorders) | 2 | 1
Abdominal Pain (Gastrointestinal disorders) | 6 | 3
Abdominal Pain (Upper) (Gastrointestinal disorders) | 9 | 2
Acne (Skin and subcutaneous tissue disorders) | 1 | 2
Activated Partial Thromboplastin Time Prolonged (Investigations) | 3 | 4
Alanine Aminotransferase Decreased (Investigations) | 0 | 2
Alanine Aminotransferase Increased (Investigations) | 5 | 5
Anxiety (Psychiatric disorders) | 10 | 11
Aphthous Stomatitis (Gastrointestinal disorders) | 2 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 4 | 3
Arthropod Bite (Injury, poisoning and procedural complications) | 2 | 1
Aspartate Aminotransferase Increased (Investigations) | 5 | 4
Blood Albumin Decreased (Investigations) | 7 | 7
Blood Alkaline Phosphatase Increased (Investigations) | 3 | 3
Blood Bicarbonate Decreased (Investigations) | 3 | 1
Blood Calcium Decreased (Investigations) | 1 | 3
Blood Calcium Increased (Investigations) | 2 | 0
Blood Creatinine Increased (Investigations) | 4 | 2
Blood Potassium Decreased (Investigations) | 0 | 2
Blood Sodium Decreased (Investigations) | 4 | 2
Blood Urea Increased (Investigations) | 2 | 0
Carbon Dioxide Abnormal (Investigations) | 2 | 0
Cardiac Murmur (Investigations) | 0 | 2
Catheter Related Complication (General disorders) | 3 | 1
Catheter Site Pain (General disorders) | 3 | 0
Catheter Site Rash (General disorders) | 3 | 1
Chills (General disorders) | 1 | 3
Conjunctivitis (Eye disorders) | 2 | 1
Constipation (Gastrointestinal disorders) | 2 | 0
Contusion (Injury, poisoning and procedural complications) | 1 | 4
Cough (Respiratory, thoracic and mediastinal disorders) | 4 | 4
Cytokine Release Syndrome (Immune system disorders) | 2 | 1
Diarrhea (Gastrointestinal disorders) | 6 | 3
Dizziness (Nervous system disorders) | 5 | 4
Dry Skin (Skin and subcutaneous tissue disorders) | 1 | 4
Dysmenorrhea (Reproductive system and breast disorders) | 0 | 2
Edema Peripheral (General disorders) | 0 | 3
Erythema (Skin and subcutaneous tissue disorders) | 2 | 1
Excoriation (Injury, poisoning and procedural complications) | 4 | 2
Fatigue (General disorders) | 3 | 8
Gamma-glutamyltransferase Increased (Investigations) | 2 | 1
Glycosylated Hemoglobin Increased (Investigations) | 2 | 3
Headache (Nervous system disorders) | 20 | 15
Hematuria (Renal and urinary disorders) | 2 | 0
Hemoglobin Decreased (Investigations) | 7 | 10
Hyperglycemia (Metabolism and nutrition disorders) | 2 | 2
Hypocalcemia (Metabolism and nutrition disorders) | 3 | 3
Hypoglycemia (Metabolism and nutrition disorders) | 3 | 6
Hyponatremia (Metabolism and nutrition disorders) | 2 | 0
Hypotension (Vascular disorders) | 3 | 2
Influenza Like Illness (General disorders) | 7 | 4/33
International Normalized Ratio Increased (Investigations) | 4 | 2/33
Ketonuria (Renal and urinary disorders) | 3 | 0/33
Laboratory Test Abnormal (Investigations) | 3 | 1/33
Leukopenia (Blood and lymphatic system disorders) | 9 | 10/33
Lipohypertrophy (Skin and subcutaneous tissue disorders) | 1 | 3/33
Lymphocyte Count Decreased (Investigations) | 0 | 5/33
Lymphocyte Count Increased (Investigations) | 2 | 0/33
Lymphopenia (Blood and lymphatic system disorders) | 10 | 15/33
Mean Cell Hemoglobin Increased (Investigations) | 2 | 0/33
Musculoskeletal Pain (Musculoskeletal and connective tissue disorders) | 0 | 3/33
Myalgia (Musculoskeletal and connective tissue disorders) | 2 | 0/33
Nasal Congestion (Respiratory, thoracic and mediastinal disorders) | 2 | 5/33
Nasopharyngitis (Infections and infestations) | 4 | 2/33
Nausea (Gastrointestinal disorders) | 11 | 14/33
Neck Pain (Musculoskeletal and connective tissue disorders) | 2 | 0/33
Neutropenia (Blood and lymphatic system disorders) | 7 | 7/33
Nodule (General disorders) | 2 | 0/33
Oral Pain (Gastrointestinal disorders) | 3 | 2/33
Pain (General disorders) | 2 | 1/33
Pain in Extremity (Musculoskeletal and connective tissue disorders) | 4 | 5/33
Petechiae (Skin and subcutaneous tissue disorders) | 2 | 0/33
Pharyngitis Streptococcal (Infections and infestations) | 0 | 2/33
Pharyngolaryngeal Pain (Respiratory, thoracic and mediastinal disorders) | 6 | 6/33
Platelet Count Decreased (Investigations) | 1 | 6/33
Protein Total Decreased (Investigations) | 3 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 9 | 11
Pyrexia (General disorders) | 6 | 8
Rash (Skin and subcutaneous tissue disorders) | 16 | 18
Rash Generalized (Skin and subcutaneous tissue disorders) | 0 | 4
Rash Papular (Skin and subcutaneous tissue disorders) | 2 | 3
Red Blood Cell Count Decreased (Investigations) | 2 | 0
Rhinitis Allergic (Respiratory, thoracic and mediastinal disorders) | 5 | 2
Skin Disorder (Skin and subcutaneous tissue disorders) | 0 | 2
Skin Exfoliation (Skin and subcutaneous tissue disorders) | 4 | 6
Skin Papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 1
Tachycardia (Cardiac disorders) | 2 | 3
Upper Respiratory Tract Infection (Infections and infestations) | 7 | 10
Urticaria (Skin and subcutaneous tissue disorders) | 2 | 2
Vomiting (Gastrointestinal disorders) | 12 | 6
White Blood Cell Count Decreased (Investigations) | 0 | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes